CLINICAL TRIAL: NCT03757234
Title: A Randomized, Double-Blinded, Adaptive Phase 2 Study to Evaluate the Safety and Efficacy of iv or iv/po Omadacycline and iv/po Levofloxacin in the Treatment of Adults With Acute Pyelonephritis.
Brief Title: IV or IV/PO Omadacycline vs. IV/PO Levofloxacin for the Treatment of Acute Pyelonephritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Paratek Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PTK0796-AP-17202
Record Dates: First submitted 2018-11-27; First posted 2018-11-28 (Actual); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Acute Pyelonephritis
MeSH Terms: interventions — omadacycline; Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Omadacycline 200 iv/200 iv (Experimental): On Day 1, participants received omadacycline 200 milligrams intravenously (iv). On Days 2 through 7, participants continued to receive omadacycline 200 milligrams iv. All doses were administered once-per-day and iv doses were administered in 150 milliliters of normal saline as continuous infusions over 90 minutes.
  Interventions: Drug: Omadacycline
- Omadacycline 200 iv/100 iv (Experimental): On Day 1, participants received omadacycline 200 milligrams iv. On Days 2 through 7, participants received omadacycline 100 milligrams iv. All doses were administered once-per-day and iv doses were administered in 150 milliliters of normal saline as continuous infusions over 90 minutes.
  Interventions: Drug: Omadacycline
- Omadacycline 200 iv/300 po or 100 iv (Experimental): On Day 1, participants received omadacycline 200 milligrams iv. On Days 2 through 7, participants received omadacycline 100 milligrams iv or omadacycline 300 milligrams per oral (po). All doses were administered once-per-day and iv doses were administered in 150 milliliters of normal saline as continuous infusions over 90 minutes. All oral doses were taken in a fasted state.
  Interventions: Drug: Omadacycline
- Omadacycline 200 iv/450 po or 100 iv (Experimental): On Day 1, participants received omadacycline 200 milligrams iv. On Days 2 through 7, participants received omadacycline 100 milligrams iv or omadacycline 450 milligrams po. All doses were administered once-per-day and iv doses were administered in 150 milliliters of normal saline as continuous infusions over 90 minutes. All oral doses were taken in a fasted state.
  Interventions: Drug: Omadacycline
- Levofloxacin 750 iv/750 po or iv (Active Comparator): On Day 1, participants received levofloxacin 750 milligrams iv. On Days 2 through 7, participants received levofloxacin 750 milligrams iv or levofloxacin 750 milligrams po. All doses were administered once-per-day and iv doses were administered in 150 milliliters of normal saline as continuous infusions over 90 minutes. All oral doses were taken in a fasted state.
  Interventions: Drug: Levofloxacin

INTERVENTIONS:
Drug: Omadacycline — po tablets
  Other Names: Nuzyra
  Arms: Omadacycline 200 iv/300 po or 100 iv; Omadacycline 200 iv/450 po or 100 iv
Drug: Levofloxacin — iv solution/po tablets
  Other Names: Levaquin
  Arms: Levofloxacin 750 iv/750 po or iv
Drug: Omadacycline — iv solution
  Other Names: Nuzyra
  Arms: Omadacycline 200 iv/100 iv; Omadacycline 200 iv/200 iv; Omadacycline 200 iv/300 po or 100 iv; Omadacycline 200 iv/450 po or 100 iv

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of intravenous (iv) or iv/per oral (po) omadacycline as compared to iv or iv/po levofloxacin in the treatment of female adults with acute pyelonephritis.

DETAILED DESCRIPTION:
This was a randomized (1:1:1:1:1), double-blind, double-dummy, adaptive designed, Phase 2 study. Based on review of the efficacy and microbiology data, the DMC modified the randomization algorithm, and no further participants were enrolled in the following treatment arms after May 2019: the omadacycline 200 iv/100 iv, omadacycline 200 iv/300 po or 100 iv, and omadacycline 200 iv/450 po or 100 iv arms. After this change, participants were randomized in a 1:1 ratio to either the omadacycline 200 iv/200 iv or levofloxacin arms.

ELIGIBILITY:
Inclusion Criteria:

* Female participants, age 18-65 years who have signed the informed consent form
* Must have a qualifying acute pyelonephritis
* Participants must not be pregnant at the time of enrollment
* Must agree to a reliable method of birth control during the study and for 30 days following the last dose of study drug
* Must be able to comply with all of the requirements of the study

Exclusion Criteria:

* Males
* Symptoms of acute pyelonephritis present for longer 7 days prior to randomization
* Infections that require antibacterial treatment for greater than 14 days
* Evidence of suspected non-renal source of infections, vaginitis, or sexually transmitted infection
* Evidence of significant immunological disease
* Evidence of liver impairment or disease
* Evidence of unstable cardiac disease
* Severe renal disease or requirement for dialysis
* Evidence of septic shock
* Has a history of hypersensitivity or allergic reaction to any tetracycline or to levofloxacin
* Has received an investigational drug within the past 30 days
* Participants who are pregnant or nursing
* Unable or unwilling to comply with the protocol requirements

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 201 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-07-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- Georgia (4):
  - Site 201, Tbilisi
  - Site 202, Tbilisi
  - Site 203, Tbilisi
  - Site 204, Tbilisi
- Latvia (5):
  - Site 301, Daugavpils
  - Site 304, Liepāja
  - Site 305, Rēzekne
  - Site 302, Riga
  - Site 303, Valmiera
- Russia (15):
  - Site 409, Krasnoyarsk
  - Site 408, Moscow
  - Site 410, Moscow
  - Site 415, Penza
  - Site 407, Rostov-on-Don
  - Site 405, Rostov-on-Don
  - Site 411, Saint Petersburg
  - Site 406, Saint Petersburg
  - Site 402, Saint Petersburg
  - Site 412, Saint Petersburg
  - Site 403, Saint Petersburg
  - Site 414, Saint Petersburg
  - Site 401, Saint Petersburg
  - Site 404, Saint Petersburg
  - Site 413, Smolensk
- Ukraine (7):
  - Site 502, Chernivtsi
  - Site 506, Dnipro
  - Site 505, Kharkiv
  - Site 504, Kyiv
  - Site 503, Kyiv
  - Site 501, Lviv
  - Site 507, Zaporizhzhia

RESULTS

PARTICIPANT FLOW:
Groups:
- Omadacycline 200 iv/300 po or 100 iv: On Day 1, participants received omadacycline 200 milligrams iv. On Days 2 through 7, participants received omadacycline 100 milligrams iv or omadacycline 300 milligrams po. All doses were administered once-per-day and iv doses were administered in 150 milliliters of normal saline as continuous infusions over 90 minutes. All oral doses were taken in a fasted state.
Period: Overall Study
Arm/Group | Omadacycline 200 iv/200 iv | Omadacycline 200 iv/100 iv | Omadacycline 200 iv/300 po or 100 iv | Omadacycline 200 iv/450 po or 100 iv | Levofloxacin 750 iv/750 po or iv
Started | 75 | 18 | 17 | 17 | 74
Completed PTE Visit | 72 | 16 | 17 | 16 | 71
Completed | 72 | 16 | 17 | 16 | 70
Not Completed | 3 | 2 | 0 | 1 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 1 | 2
Not completed — Other | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population consisted of all randomized participants regardless of whether or not the participant received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Omadacycline 200 iv/200 iv | Omadacycline 200 iv/100 iv | Omadacycline 200 iv/300 po or 100 iv | Omadacycline 200 iv/450 po or 100 iv | Levofloxacin 750 iv/750 po or iv | Total
Number analyzed (Participants) | 75 | 18 | 17 | 17 | 74 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (14.97) | 33.9 (14.48) | 37.1 (15.97) | 38.2 (17.66) | 38.8 (14.74) | 37.9 (15.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 18 | 17 | 17 | 74 | 201
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 74 | 18 | 17 | 17 | 74 | 200
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 74 | 18 | 17 | 17 | 74 | 200
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Investigator Assessment of Clinical Response at the Post Therapy Evaluation (PTE) Visit (ITT Population)
Description: Clinical response was determined by the investigator at the PTE visit by assessing whether or not the participant met the clinical outcome of Clinical Success, Clinical Failure, or Indeterminate. Clinical Success was defined as the complete resolution or significant improvement of the baseline AP signs and symptoms at the PTE visit such that no additional antimicrobial therapy is required for the current infection. Clinical Failure was defined as no apparent response to therapy or persistence of signs and symptoms of infection or reappearance of signs and symptoms at or before the PTE visit such that use of additional systemic antimicrobial therapy for the current infection was required or death at or before the PTE visit. The clinical outcome was deemed as Indeterminate when the PTE visit was not completed.
Time Frame: Day 21 (A PTE occurred on Day 21 ± 2 days after the participant's first dose of study drug).
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 200 iv/200 iv | Omadacycline 200 iv/100 iv | Omadacycline 200 iv/300 po or 100 iv | Omadacycline 200 iv/450 po or 100 iv | Levofloxacin 750 iv/750 po or iv
Number analyzed (Participants) | 75 | 18 | 17 | 17 | 74
Participants
  Clinical Success | 68 | 15 | 15 | 16 | 69
  Clinical Failure | 5 | 1 | 2 | 0 | 1
  Indeterminate | 2 | 2 | 0 | 1 | 4
Statistical Analysis 1: Comparison: Omadacycline 200 iv/200 iv vs Levofloxacin 750 iv/750 po or iv; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -2.6, 95% CI 2-sided [-12.4 to 6.9] — Point estimate and exact 95% confidence intervals for difference from levofloxacin (omadacycline minus levofloxacin) in clinical success rate was estimated
Statistical Analysis 2: Comparison: Omadacycline 200 iv/100 iv vs Levofloxacin 750 iv/750 po or iv; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -9.9, 95% CI 2-sided [-34.8 to 5.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Omadacycline 200 iv/300 po or 100 iv vs Levofloxacin 750 iv/750 po or iv; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -5.0, 95% CI 2-sided [-30.6 to 8.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Omadacycline 200 iv/450 po or 100 iv vs Levofloxacin 750 iv/750 po or iv; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment Difference = 0.9, 95% CI 2-sided [-22.4 to 11.8] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Number of Participants With a Microbiological Response at the PTE Visit (Micro-ITT Population)
Description: Microbiological response was determined programmatically at the PTE visit by assessing whether or not the participant met the microbiological outcome of 'Success', 'Failure', or 'Indeterminate'. Participants were considered to have a microbiological response of 'Success' if the outcomes of each baseline pathogens were eradication at the PTE visit. Participants were considered to have a microbiological response of 'Failure' if the outcome for any pathogen was persistence. Participants were considered to have a microbiological response of 'Indeterminate', if the outcome of at least 1 baseline pathogen was indeterminate and there was no outcome of persistence for any baseline pathogen.
Time Frame: Day 21 (A PTE occurred on Day 21 ± 2 days after the participant's first dose of study drug).
Population: The micro-ITT population consisted of participants in the ITT population who had an appropriately collected pretreatment baseline urine culture with at least 1 uropathogen at ≥10^5 colony forming unit (CFU)/mL and not more than 2 bacterial isolates at any colony count.
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 200 iv/200 iv | Omadacycline 200 iv/100 iv | Omadacycline 200 iv/300 po or 100 iv | Omadacycline 200 iv/450 po or 100 iv | Levofloxacin 750 iv/750 po or iv
Number analyzed (Participants) | 46 | 11 | 14 | 13 | 52
Participants
  Clinical Success | 32 | 3 | 9 | 5 | 39
  Clinical Failure | 13 | 7 | 5 | 7 | 11
  Indeterminate | 1 | 1 | 0 | 1 | 2
Statistical Analysis 1: Comparison: Omadacycline 200 iv/200 iv vs Levofloxacin 750 iv/750 po or iv; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -5.4, 95% CI 2-sided [-23.6 to 12.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Omadacycline 200 iv/100 iv vs Levofloxacin 750 iv/750 po or iv; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -47.7, 95% CI 2-sided [-71.3 to -6.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Omadacycline 200 iv/300 po or 100 iv vs Levofloxacin 750 iv/750 po or iv; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -10.7, 95% CI 2-sided [-40.8 to 15.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Omadacycline 200 iv/450 po or 100 iv vs Levofloxacin 750 iv/750 po or iv; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -36.5, 95% CI 2-sided [-62.6 to -1.1] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Number of Participants With Resolution of All AP Signs and Clinical Symptoms at PTE Visit (ITT Population)
Description: Participants recorded their assessments using the Modified Patient Symptom Assessment Questionnaire (mPSAQ), a 6-item questionnaire that assessed the levels of 'severity' and 'bothersomeness' for six pyelonephritis signs and symptoms. The sub-scale responses were recorded as 'did not have', 'mild', 'moderate', and 'severe' for 'severity'; and 'not at all', 'a little', 'moderately', and 'a lot' for 'bothersomeness', both scored 0-3. Total scores were calculated by summing the non-missing scores of the 6 items, divided by the number of non-missing items, and then multiplied by 6. For each sub-scale, the total score ranged from 0 (least Severe/ least bothersome) and 18 (worst severity/most bothersome). Number of participants with resolution of all symptoms, without occurrence of new symptoms is reported. Resolution was defined as absence of all baseline symptoms.
Time Frame: Day 21 (A PTE occurred on Day 21 ± 2 days after the participant's first dose of study drug).
Population: The ITT population consisted of all randomized participants regardless of whether or not the participant received study drug. Participants who completed the PTE visit with evaluable data were analyzed for this end point.
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 200 iv/200 iv | Omadacycline 200 iv/100 iv | Omadacycline 200 iv/300 po or 100 iv | Omadacycline 200 iv/450 po or 100 iv | Levofloxacin 750 iv/750 po or iv
Number analyzed (Participants) | 64 | 16 | 16 | 16 | 66
Participants | 51 | 15 | 14 | 13 | 54

4. Primary Outcome: Number of Participants With No Worsening and Absence of New AP Signs and Clinical Symptoms at PTE Visit (ITT Population)
Description: Participants recorded their assessments using the mPSAQ, a 6-item questionnaire that assessed the levels of 'severity' and 'bothersomeness' for six pyelonephritis signs and symptoms. The sub-scale responses were recorded as 'did not have', 'mild', 'moderate', and 'severe' for 'severity'; and 'not at all', 'a little', 'moderately', and 'a lot' for 'bothersomeness', both scored 0-3. Total scores were calculated by summing the non-missing scores of the 6 items, divided by the number of non-missing items, and then multiplied by 6. For each sub-scale, the total score ranged from 0 (least Severe/ least bothersome) and 18 (worst severity/most bothersome). Number of participants with no worsening and absence of AP signs and clinical symptoms is reported. No worsening meant that each question score is same or better at post baseline.
Time Frame: Day 21 (A PTE occurred on Day 21 ± 2 days after the participant's first dose of study drug).
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 200 iv/200 iv | Omadacycline 200 iv/100 iv | Omadacycline 200 iv/300 po or 100 iv | Omadacycline 200 iv/450 po or 100 iv | Levofloxacin 750 iv/750 po or iv
Number analyzed (Participants) | 64 | 16 | 16 | 16 | 66
Participants | 62 | 16 | 16 | 15 | 65

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events and Serious Adverse Events
Description: An adverse event is any untoward, undesired, or unplanned event in the form of signs, symptoms, disease, or laboratory or physiologic observations occurring in a person given a study drug or in a clinical study. A treatment-emergent adverse event was defined as any adverse event that newly appeared, increased in frequency, or worsened in severity on or after the initiation of the study drug.
Time Frame: up to approximately 28 days
Population: The Safety population consisted of all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 200 iv/200 iv | Omadacycline 200 iv/100 iv | Omadacycline 200 iv/300 po or 100 iv | Omadacycline 200 iv/450 po or 100 iv | Levofloxacin 750 iv/750 po or iv
Number analyzed (Participants) | 75 | 18 | 17 | 17 | 74
Participants
  Treatment Emergent Adverse Events | 23 | 6 | 9 | 8 | 24
  Treatment Emergent Serious Adverse Events | 0 | 0 | 2 | 2 | 2

ADVERSE EVENTS:
Time Frame: Up to approximately 28 days
Description: The Safety Population consisted of all randomized participants who received at least one dose of study drug.
Arm/Group | Omadacycline 200 iv/200 iv | Omadacycline 200 iv/100 iv | Omadacycline 200 iv/300 po or 100 iv | Omadacycline 200 iv/450 po or 100 iv | Levofloxacin 750 iv/750 po or iv
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/18 | 0/17 | 0/17 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/18 | 2/17 | 2/17 | 2/74
Other Adverse Events (participants affected / at risk) | 21/75 | 6/18 | 7/17 | 8/17 | 16/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omadacycline 200 iv/200 iv (N=75) | Omadacycline 200 iv/100 iv (N=18) | Omadacycline 200 iv/300 po or 100 iv (N=17) | Omadacycline 200 iv/450 po or 100 iv (N=17) | Levofloxacin 750 iv/750 po or iv (N=74)
Renal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omadacycline 200 iv/200 iv (N=75) | Omadacycline 200 iv/100 iv (N=18) | Omadacycline 200 iv/300 po or 100 iv (N=17) | Omadacycline 200 iv/450 po or 100 iv (N=17) | Levofloxacin 750 iv/750 po or iv (N=74)
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 5
Nausea (Gastrointestinal disorders) | 3 | 0 | 0 | 4 | 5
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Asthenia (General disorders) | 2 | 0 | 0 | 0 | 1
Hyperthermia (General disorders) | 0 | 1 | 0 | 0 | 0
Asymptomatic bacteriuria (Infections and infestations) | 3 | 2 | 2 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Viral rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 8 | 0 | 2 | 3 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1

LIMITATIONS AND CAVEATS:
In May 2019, the DMC modified the randomization algorithm based on their review of the data. After this change, participants were randomized in a 1:1 ratio to either the omadacycline 200 iv/200 iv or levofloxacin arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the Principal Investigator is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor can request changes to the communication and require the removal of confidential information.

DOCUMENTS (2):
  • Study Protocol (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/34/NCT03757234/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-04): https://cdn.clinicaltrials.gov/large-docs/34/NCT03757234/SAP_001.pdf